CLINICAL TRIAL: NCT00169000
Title: Phase I Study of a Novel Schedule of Capecitabine and Docetaxel in Patients With Advanced Solid Tumors
Brief Title: Safety Study of a New Schedule of Capecitabine and Docetaxel to Treat Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Gary N. Schwartz, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0139
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; capecitabine; docetaxel; pharmacokinetic/pharmacodynamic; bcl-2; bax
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Capecitabine and Docetaxel (Experimental): Escalating doses of capecitabine days 1-14 with a fixed dose of docetaxel on Day 8 of a 21 day cycle
  Interventions: Drug: Capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Capecitabine — Capecitabine at the following dose levels for 14 days every 21 days, beginning with dose level 1
  Dose level -2 600 mg/m2 po BID
  Dose level -1 700 mg/m2 po BID
  Dose level 1 825 mg/m2 po BID
  Dose level 2 1000 mg/m2 po BID
  Other Names: Xeloda
Drug: Docetaxel — 75 mg/m2 over one hour on day 8 of each cycle
  Other Names: Taxotere

SUMMARY:
The combination of capecitabine and docetaxel is given to treat several different types of cancer. Capecitabine is usually given by mouth for 14 days, and docetaxel is given IV on the first day of capecitabine. The effects of changes in the schedule of the combination of docetaxel and capecitabine has been examined in human breast cancer cells. A capecitabine by-product was given orally to breast cancer-bearing animals for 14 consecutive days. Docetaxel was given IV at a variety of times between days 1 and 15. The greatest reductions in the volume of the cancer were seen when animals were treated with docetaxel between days 6 and 10. In two other breast cancer models, the maximal degree of delay in growth of the tumors was achieved when the animals were treated with docetaxel on day 8 of a 14 day course of capecitabine. The extent of tumor response was not explained by changes in tumor levels of the enzyme thymidine phosphorylase, which is thought to be the mechanism behind the interaction of capecitabine and docetaxel. In the breast cancer cells, capecitabine increases the level of proteins which promote death of cancer cells, and it inhibits the levels of proteins which block death of cancer cells.

Our hypothesis is that capecitabine and docetaxel interact with each other, because capecitabine primes the pro-death machinery of the cell by increasing the ratio of death-promoting proteins to death-inhibiting proteins. Cells are more susceptible to killing by docetaxel when the pro-death machinery is activated by capecitabine.

This is a safety study to find the highest dose of capecitabine that can be given safely for 14 days, in combination with docetaxel given at a fixed dose on day 8. Once this dose of capecitabine has been determined, an additional nine patients with tumors that can be biopsied will be treated at this dose, and levels of capecitabine, its byproducts, and docetaxel will be measured in the bloodstream. Biopsies of tumors will also be taken before and after the docetaxel is given, and the levels of pro-death and anti-death proteins will be measured.

DETAILED DESCRIPTION:
This is a phase I study using an accelerated titration design to determine the maximum tolerated dose (MTD) of capecitabine given orally on a BID schedule from days 1-14, in combination with docetaxel given at a fixed dose of 75 mg/m2 IV on day 8. Once the MTD of capecitabine has been determined, an additional nine patients with accessible tumors will be treated at the MTD. Pharmacokinetics of plasma capecitabine, 5-FU, 5'-deoxy-5-fluorouridine, and docetaxel will be assayed in these nine patients, and tumor biopsies will be taken to assess Bax:Bcl-2 ratios and Bcl-2 phosphorylation at several time points. The primary aim of this study will be to determine the maximum tolerated dose and dose limiting toxicities of capecitabine when given with a fixed dose of docetaxel on day 8 of a 21 day schedule. Secondary aims will include assessment of the pharmacokinetics of capecitabine and docetaxel on this schedule, and determination of intratumoral Bax:Bcl-2, Bcl-2 phosphorylation, and DPD expression, and correlation with clinical toxicities and antitumor response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically or cytologically proven metastatic solid tumor.
* Patients with measurable disease or an evaluable bone lesion that will not undergo biopsy.
* Patients treated within the additional cohort at MTD will have metastatic breast cancer with a site of disease that is amenable to percutaneous FNA and must be willing to undergo serial FNA biopsies of their primary tumor.
* Age > 18 years.
* Life expectancy of at least 6 months.
* ECOG performance status 0-2.
* Adequate hematologic, hepatic, and renal function
* Patients must have an intact upper gastrointestinal tract, be able to swallow tablets, and not have a malabsorption syndrome.

Exclusion Criteria:

* No significant uncontrolled infectious or cardiovascular disease, or a myocardial infarction within the prior 12 months.
* No prior organ allograft.
* No prior treatment with capecitabine or with docetaxel.
* No prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
* No concurrent antacid therapy is allowed.
* No other significant medical/surgical diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-01; Primary Completion 2005-09 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose, and dose limiting toxicity of capecitabine when given daily for 14 days with docetaxel given on day 8 of a 21 day cycle | 3 weeks

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of capecitabine, 5-fluorouracil, and 5'-deoxy-5-fluorouridine following administration of docetaxel on day 8. | 9 days
To determine the expression of Bax, Bcl-2, and phosphorylated Bcl-2 at baseline and again on days 8 and 9 of capecitabine when given at the MTD | 9 days
To define pharmacodynamic relationships between observed changes in dihydropyrimidine dehydrogenase (DPD) and altered expression of Bax and Bcl-2 with clinical toxicities and antitumor response | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Schwartz, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States